CLINICAL TRIAL: NCT04822558
Title: The Relevance of a 3D Multisegment Foot Model in Predicting and Determining the Clinical Outcome After Ankle and Hindfoot Reconstruction Procedures
Brief Title: 3D Multisegment Foot Model Used for the Clinical Outcome After Ankle and Hindfoot Reconstruction
Acronym: 3D-MFM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S55070
Record Dates: First submitted 2021-03-17; First posted 2021-03-30 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Ankle and Hindfoot Alterations
Keywords: 3D multisegment foot model
MeSH Terms: interventions — Gait Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ankle and hindfoot reconstruction surgery (Other): Patients who underwent an ankle- or hindfoot reconstruction surgery
  Interventions: Other: Plantar pressure measurement; Other: Gait analysis; Procedure: Ankle and hindfoot reconstruction surgery

INTERVENTIONS:
Other: Plantar pressure measurement — Biomechanical and clinical evaluation of the reconstructive procedures of ankle and hindfoot using a 3D multisegment foot model
Other: Gait analysis — Biomechanical and clinical evaluation of the reconstructive procedures of ankle and hindfoot using a 3D multisegment foot model
Procedure: Ankle and hindfoot reconstruction surgery — Ankle and hindfoot reconstruction surgery

SUMMARY:
Most symptomatic pathologies of the ankle and hindfoot are determined by biomechanical alterations of this anatomical region. Surgical treatment of these pathologies is therefore aimed at improving the inferior biomechanical condition, and it can be expected that an improvement of the biomechanical parameters grossly parallels the targeted clinical improvement.

3D Multisegment Foot Models have been developed and validated to determine the clinical outcome. Such a validated 3D Multisegment Foot Model is now standard available in the gaitlab of UZ Leuven making it possible to study a huge amount of biomechanical parameters within the foot & ankle region itself.

DETAILED DESCRIPTION:
Most symptomatic pathologies of the ankle and hindfoot are determined by biomechanical alterations of this anatomical region. Surgical treatment of these pathologies is therefore aimed at improving the inferior biomechanical condition, and it can be expected that an improvement of the biomechanical parameters grossly parallels the targeted clinical improvement.

Unfortunately, in the past, biomechanical examination of the lower limb and foot consisted of two distinct study protocols: gaitlab and plantar pressure measurements.

First, these two study protocols were acquired completely independently. Therefore, it proved to be very hard to compare the results and get insight in the way altered biomechanics caused or continued to cause abnormal plantar pressure distributions. However, recently it was possible to integrate these two modalities, especially concerning the timing of the events, what makes it possible to reliably link the observed findings.

Second, virtually all gaitlab models considered the foot & ankle region as one single segment, making it impossible to evaluate any biomechanical parameter within the targeted region. 3D Multisegment Foot Models have been developed and validated since the beginning of this century. Such a validated 3D Multisegment Foot Model is now standard available in the gaitlab of UZ Leuven making it possible to study a huge amount of biomechanical parameters within the foot & ankle region itself.

Furthermore, only a paucity of information is available if the observed clinical changes are indeed paralleled by an equally directed biomechanical change.

Historically, all patients at the Foot & Ankle unit of UZ Leuven performed a pre- and 1 year post-operative plantar pressure measurement to get better insight in their clinical condition. As stated before, the usefulness of this single testing method was limited. Recently the Advanced Clinical Examination Platform that integrates both plantar pressure measurement and full 3D MFM-gaitlab has been implemented in the Movement Analysis Laboratory of our institution. Currently a transition to routinely perform such an examination is finished. Therefore a completely new era of research concerning the biomechanical evaluation itself and clinical results of the reconstructive procedures of ankle and hindfoot has started.

ELIGIBILITY:
Inclusion Criteria:

* Being routinely scheduled for a reconstructive surgical procedure for the following indications or involving the following type of procedure:

  1. Any reconstructive procedure for Pes Planus, Pes Plano-valgus, or Posterior Tibial Tendon Dysfunction
  2. Tibio-talar arthrodesis or prosthesis
  3. Sub-talar -and/or (partial) Chopart - and/or Triple arthrodesis
  4. Pantalar arthrodesis with or without inclusion of the Chopart joint

     Exclusion Criteria:
* Age under 18
* Need of tools (eg walker or crutches) to walk less than 100m
* Inability to walk less than 100 m anyway
* Differences in leg length exceeding 3 cm (measured clinically)
* Extreme in-or outtoeing
* Subjects with BMI > 27.5 require very careful further consideration whether or not the obesity prevents the accurate palpation of anatomical landmarks necessary prior to marker placement. This will be judged on an individual basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Gaitlab parameters | Pre-operative and at 1 year
  To determine the correlation between the observed changes in gaitlab parameters and the observed changes at plantar pressure measurement and to determine if a clear correlation can be determined, comparing the pre- and post-operative results 3D multisegment foot model testing and clinical outcome

SECONDARY OUTCOMES:
3D motion analysis: Gaitlab parameters to determine biomechanical parameters | Pre-operative and at 1 year
  To determine which biomechanical parameter is the driving force for specific clinical observations using a 3D multisegment foot model
Foot Function Index (FFI) | Pre-operative, at 6 months and at 1 year
  To measure the impact of foot pathology on function in terms of pain, disability and activity restriction
Short Form 36 Health Survey Questionnaire (SF-36) | Pre-operative, at 6 months and at 1 year
  To indicate the health status and pain scales
Visual Analog Scale (VAS) | Pre-operative, at 6 months and at 1 year
  To determine the pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Matricali, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No